CLINICAL TRIAL: NCT05503303
Title: Clinical Characteristics in Adults With Type 1 Diabetes, Metabolic Syndrome and Insulin Resistance
Brief Title: T1D, Metabolic Syndrome and Insulin Resistance
Status: Completed | Type: Observational
Sponsor: Universidad Juárez Autónoma de Tabasco (Other)
Responsible Party: Principal Investigator, ISELA ESTHER JUAREZ-ROJOP Ph.D., Full-Time Investigator Professor, Universidad Juárez Autónoma de Tabasco
Other Study IDs: T1D-DACS2022
Record Dates: First submitted 2022-08-13; First posted 2022-08-16 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Type 1 Diabetes; Metabolic Syndrome; Insulin Resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Metabolic Syndrome; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with type 1 diabetes (T1D) and metabolic syndrome (MS) require high doses of insulin to achieve a glycemic control, due to insulin resistance (IR). The investigators identified the presence of metabolic syndrome and insulin resistance in patients with T1D in a population of southeast Mexico.

The sampled population was recruited from the Diabetes Clinic of the Regional Hospital of High Specialty "Dr. Gustavo A. Rovirosa Pérez"; from August 2021 to February 2022, graduated physicians interviewed patients previously diagnosed with T1D. This study included patients older than 18 years and at least six months after being diagnosed with T1D. The interviewers excluded patients who did not attend regular consultations and those who did not agree to participate or to give a blood sample. A diabetologist evaluated and diagnosed all patients based on the World Health Organization (WHO) criteria.

Fasting glucose, total cholesterol, HDL cholesterol, LDL cholesterol, and triacylglycerols were determined in blood serum using a Clinical Chemistry System from Random Access Diagnostics. The reasearch team determined glycated hemoglobin concentrations by an enzymatic immunoassay method.

ELIGIBILITY:
Inclusion Criteria:

* At least six months after being diagnosed with T1D

Exclusion Criteria:

* Did not attend regular consultations
* Did not agree to participate or to give a blood sample

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients who attend Diabetes Clinic of the Regional Hospital of High Specialty "Dr. Gustavo A. Rovirosa Pérez", previously diagnosed with type 1 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Glycated hemoglobin | March 2022
  Concentrations by an enzymatic immunoassay method
Total cholesterol, HDL cholesterol, LDL cholesterol, and triacylglycerols | March 2022
  Determined in blood serum using a Clinical Chemistry System from Random Access Diagnostics

CONTACTS AND LOCATIONS:
Locations (1):
- Isela Esther Juarez Rojop, Villahermosa, Tabasco, Mexico